CLINICAL TRIAL: NCT06955156
Title: Trilaciclib in Combination With Anti-PD-1 Antibody and Chemotherapy in the Treatment of Locally Advanced Triple-negative Breast Cancer: A Prospective, Single-arm, Multicenter Phase II Clinical Study
Brief Title: Trilaciclib Combined With Anti-PD-1 Antibody and Chemotherapy in the Treatment of Locally Advanced TNBC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: QIAO LI (Other)
Responsible Party: Sponsor-Investigator, QIAO LI, Chief physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Trila-CN-BC-01
Record Dates: First submitted 2024-08-03; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-07

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — trilaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Trilaciclib + Anti-PD-1 Antibody + Chemotherapy
  Interventions: Drug: Trilaciclib

INTERVENTIONS:
Drug: Trilaciclib — trilaciclib 240mg/m2 ivgtt d1 Q3w; anti-PD-1 antibody 200mg ivgtt d1 Q3w; Paclitaxel-albumin 250mg/m2 ivgtt d1 Q3w or 125mg/m2 ivgtt d1,d8 Q3w; carboplatin AUC=5 ivgtt d1 Q3w; Review every 2 cycles until the best efficacy or intolerable toxicity, usually 6-8 cycles;
  Other Names: Cosela

SUMMARY:
Trilaciclib is a highly potent, selective, and reversible CDK4/6 inhibitor that protects bone marrow by protecting hematopoietic stem cells and progenitor cells (HSPCs) during systemic chemotherapy. The proliferation and differentiation of HSPCs are highly dependent on the CDK4/6 signaling pathway, and when exposed to the appropriate dose of treacilil, they will be blocked in the G1 phase of the cell cycle, thus avoiding the killing of cell cycle-specific chemotherapy drugs. This is an open, single-arm, multicenter Phase II clinical study. Newly diagnosed TNBC patients with T1c N1-2 or T2-4 N0-2 will be screened according to the inclusion criteria. Fifty patients meeting the inclusion criteria will sign informed consent letters and receive neoadjuvant therapy with Trilaciclib + anti-PD-1 antibody + Paclitaxel-albumin + carboplatin. To evaluate the synergistic effect of Trilaciclib on bone marrow protection and anti-tumor therapy.

DETAILED DESCRIPTION:
Myelosuppression is the cause of many cancer chemotherapy-related adverse events, such as infections, sepsis, bleeding, and fatigue, resulting in delayed hospital stays or the need for treatment with hematopoietic growth factors, blood transfusions, and so on. In addition, myelosuppression usually leads to a lower dose or more extended interval of chemotherapy, which reduces the intensity of chemotherapy and affects the benefit of chemotherapy for patients.

Trilaciclib is a highly potent, selective, and reversible CDK4/6 inhibitor that protects bone marrow by protecting hematopoietic stem cells and progenitor cells (HSPCs) during systemic chemotherapy. The proliferation and differentiation of HSPCs are highly dependent on the CDK4/6 signaling pathway, and when exposed to the appropriate dose of treacilil, they will be blocked in the G1 phase of the cell cycle, thus avoiding the killing of cell cycle-specific chemotherapy drugs. This is an open, single-arm, multicenter Phase II clinical study. Newly diagnosed TNBC patients with T1c N1-2 or T2-4 N0-2 will be screened according to the inclusion criteria. Fifty patients meeting the inclusion criteria will sign informed consent letters and receive neoadjuvant therapy with Trilaciclib + anti-PD-1 antibody + Paclitaxel-albumin + carboplatin. To evaluate the synergistic effect of Trilaciclib on bone marrow protection and anti-tumor therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients fully understand and voluntarily participate in this study and sign the informed consent form.
2. Age ≥18 and ≤75 years.
3. Newly diagnosed TNBC with stage T1c N1-3 or stage T2-4 N0-3.
4. Patients scheduled to receive neoadjuvant therapy.
5. Patients have measurable lesions (non-lymph node lesions ≥10 mm in length and lymph node lesions ≥15 mm in length according to RECIST 1.1 standards).
6. No previous antitumor system therapy.
7. ECOG (Eastern Cooperative Oncology Group) performance status of 0-1.
8. Patients voluntarily joined the study with nice compliance.
9. Good organ function (no blood transfusion or growth factor support within 2 weeks before the first dose of trial medication): WBC≥3.0×10^9/L, ANC ≥1.5×10^9/L, PLT ≥75×10^9/L, Hb≥90g/L, ALP≤5×ULN, ALT≤3×ULN, AST≤3×ULN, ALB≥28 g/L, Creatinine≤1.5×ULN or Creatinine clearance ≥50 mL/min, INR≤1.5 /PT≤1.5×ULN, aPTT≤1.5×ULN (If patient is receiving anticoagulant therapy, as long as the PT INR is within the prescribed range of anticoagulants).

Exclusion Criteria:

1. Pathological diagnosis of HR+ or HER2+ breast cancer.
2. Imaging shows metastatic breast cancer.
3. Previous or current concurrent malignancy other than breast cancer.
4. Patients had any active autoimmune disease or a history of autoimmune disease (e.g., but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary vasculitis, nephritis, hyperthyroidism; Patients had vitiligo; Patients who had complete remission of asthma in childhood and without any intervention in adulthood were included; Patients with asthma requiring medical intervention with bronchodilators were not included).
5. Patients are taking immunosuppressants or systemic hormone therapy for immunosuppressive purposes (dose > 10mg/day of prednisone or other therapeutic hormone) and continued use within 2 weeks prior to enrollment.
6. Recurrence after surgery, previous local or systemic antitumor therapy.
7. Patients are known to have a prior allergy to the drug ingredient being applied.
8. Patients with poorly controlled cardiac clinical symptoms or diseases, such as (1)NYHA2 or higher heart failure, (2) unstable angina pectoris, (3) myocardial infarction within 1 year, (4) Clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention.
9. Patients with active infection or unexplained fever during screening or prior to initial treatment >38.5℃ (as determined by the investigator, the subject's fever due to the tumor can be enrolled).
10. Live vaccine was administered less than 4 weeks before or possibly during the study period
11. Patients have a known history of psychotropic substance abuse, alcohol abuse, or druggy use.
12. Patients should be excluded if, in the investigator's judgment, the subjects have other factors that may cause the study to be terminated (other severe medical conditions requiring concomitant treatment, serious laboratory abnormalities, associated family or social factors, and other circumstances that may affect the safety of the subjects or the collection of data and samples).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of ≥ grade 3 neutropenia during chemotherapy | At the end of Cycle 1 (each cycle is 21days)
  Incidence of ≥ grade 3 neutropenia during chemotherapy. (neutrophil count ≤ 1*10^9/L）

SECONDARY OUTCOMES:
event-free survival | one year after the last dose
  Time from randomization to occurrence of any event
Duration of grade 3 or 4 neutropenia in the first treatment cycle of chemotherapy (days); | From the initiation of the first dose to 28 days after the last dose
  Duration of grade 3 or 4 neutropenia in the first treatment cycle of chemotherapy (days)
The incidence of grade 3 or 4 thrombocytopenia | From the initiation of the first dose to 28 days after the last dose
  The incidence of grade 3 or 4 thrombocytopenia (Platelet<50×109/L)
The incidence of grade 3 or 4 anemia during chemotherapy treatment | From the initiation of the first dose to 28 days after the last dose
  The incidence of grade 3 or 4 anemia during chemotherapy treatment (HGB<80g/L)
Incidence of adverse events (AES) and serious adverse events (SAEs) | From the initiation of the first dose to 28 days after the last dose
  The incidence of adverse events (AES) and serious adverse events (SAEs), and the incidence of AES/SAEs leading to treatment termination
pathologic complete response (pCR) | At the end of Cycle 6-8 (each cycle is 21 days)
  Proportion of patients with no residual invasive tumor cells on pathological examination of primary breast lesions and axillary lymph node surgical specimens of all patients
Utilization rate of Granulocyte colony stimulation (G-CSF) | From the initiation of the first dose to 28 days after the last dose
  Utilization rate of Granulocyte colony stimulation (G-CSF)
All-cause chemotherapy dose reduction rate. | From the initiation of the first dose to 28 days after the last dose
  All-cause chemotherapy dose reduction rate.

CONTACTS AND LOCATIONS:
Overall Officials: Qiao Li, Principal Investigator — National Cancer Center/Cancer Hospital
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No